CLINICAL TRIAL: NCT01159054
Title: Novel Pathways to Manage Inflammation and Atherosclerosis in Dialysis Patients: Role of Nicotinic Acid
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The funding source is not going to fund this anymore. Only two subjects completed the study therefore meaningful analysis not possible.
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Kambiz Zandi-Nejad, MD, Instructor in Medicine, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010P001049
Record Dates: First submitted 2010-07-07; First posted 2010-07-09 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-05

CONDITIONS: Dialysis; Cardiovascular Disease; Atherosclerosis; Inflammation
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis; Inflammation | interventions — Niacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- This study has only one arm. (Experimental): Blood sample and scan results to be compared before and after intervention in each subject.
  Interventions: Drug: Extended Release Nicotinic Acid (Niaspan)

INTERVENTIONS:
Drug: Extended Release Nicotinic Acid (Niaspan) — Subjects will start on 500 mg per day of Niaspan for 4 weeks, then the dose will be increased to 1000 mg per day of Niaspan for 4 weeks, then the dose will be increased to 1500 mg of Niaspan per day for 4 weeks, after this subjects with weight of less than 60 kg will continue at 1500 mg per day of Niaspan for another 12 weeks whereas in subjects with weight of more than 60 kg the dose will be increased to 2000 mg of Niaspan per day which will be continued for 12 weeks.
  Other Names: Extended Release Nicotinic Acid; Niaspan

SUMMARY:
Patients with kidney failure on hemodialysis have an extremely high rate of cardiovascular disease including atherosclerotic cardiovascular disease. This, at least in part, is due to the chronic inflammatory status usually seen in these patients. Here we try to see if treatment with extended release nicotinic acid (Niaspan) can reduce their overall inflammatory burden (in general) and the atherosclerotic plaque inflammation (in particular).

ELIGIBILITY:
Inclusion Criteria:

* A signed consent form;
* Male or Female, 18 years or older;
* Diagnosed with ESRD, on maintenance hemodialysis for at least six (6) months;
* Subject must be able to understand and provide informed consent;
* No known contraindications to therapy with nicotinic acid;
* Female subjects of childbearing potential must be willing to be on an acceptable form of birth control for the duration of the study and for two month after they have stopped taking the study drug.

Exclusion Criteria:

* Any patient with a medical condition or taking any medications that would be contraindicated with the use of extended release niacin, such as active peptic ulcer disease;
* History of severe allergic reactions to the study medication;
* History of active infection or acute gouty attack within 2 weeks prior to enrollment;
* Known serological positivity for HIV, HBsAg, or HCV Ab;
* HbA1C > 9;
* Total CK of more than three times of the upper limit of normal;
* Elevation of liver function tests at time of entry (AST and/or ALT > 2 times the upper limit of normal);
* History of drug, alcohol, or chemical abuse within 6 months prior to enrollment;
* History of malignancy except adequately treated in-situ cervical carcinoma, or adequately treated basal or squamous cell carcinoma of the skin;
* History of an inflammatory disease such as SLE, rheumatoid arthritis or ulcerative colitis;
* Patients currently on pharmacological doses of nicotinic acid;
* Patients receiving chronic anti-inflammatory therapy;
* Patients with average baseline hs-CRP levels of > 20 mg/L or < 1 mg/L;
* Patients in whom FDG-PET/CT dual scans are contraindicated (e.g., pregnant patients or those with severe allergy to IV contrast; a pregnancy test will be performed in each female subject between 18 and 45 years of age prior to each scan)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kambiz ZANDI-NEJAD, MD, Principal Investigator — Brigham and Women's Hospital
Locations (3):
- United States (3):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - BWH/FH/DCI Outpatient Dialysis Unit, Boston, Massachusetts
  - DCI Dialysis Unit-Somerville, Somerville, Massachusetts

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group (One Arm Only Study): Blood sample and scan results to be compared before and after intervention in each subject.
  Extended Release Nicotinic Acid (Niaspan): Subjects will start on 500 mg per day of Niaspan for 4 weeks, then the dose will be increased to 1000 mg per day of Niaspan for 4 weeks, then the dose will be increased to 1500 mg of Niaspan per day for 4 weeks, after this subjects with weight of less than 60 kg will continue at 1500 mg per day of Niaspan for another 12 weeks whereas in subjects with weight of more than 60 kg the dose will be increased to 2000 mg of Niaspan per day which will be continued for 12 weeks.
Period: Overall Study
Arm/Group | Treatment Group (One Arm Only Study)
Started | 22
Completed | 2
Not Completed | 20

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Group (One Arm Only Study)
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 8
Age, Continuous [Mean (Full Range); unit: years] | 58.9 [25 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Changes in FDG-PET/CT Dual Scan Score
Time Frame: 6 months
Population: Analysis of images for this outcome measure was not done given than only 2 subjects had completed the study at the time of the study early termination and closure (per funding source)
Arm/Group | Treatment Group (One Arm Only Study)
Number analyzed (Participants) | 0
Value | 0

2. Primary Outcome: Changes in Hs-CRP Level
Description: Change in hs-CRP level before and after treatment in each subject
Time Frame: 6 months
Population: Only 2 subjects completed the study. Power for further analysis was not met.
Measure: Mean (Full Range); unit: mg/L
Arm/Group | Treatment Group (One Arm Only Study)
Number analyzed (Participants) | 2
mg/L
  Average Pre-Treatment | 18.465 [9.09 to 27.84]
  Average Post-Treatment | 26.395 [8.76 to 44.03]

3. Primary Outcome: Changes in IL-6 Level
Description: Change in IL-6 level before and after treatment in each subject
Time Frame: 6 months
Population: Only 2 subjects completed the study. Further analysis not done because power was not met.
Measure: Mean (Full Range); unit: pg/mL
Arm/Group | Treatment Group (One Arm Only Study)
Number analyzed (Participants) | 2
pg/mL
  Average Pre-Treatment | 5.1254 [1.962 to 8.287]
  Average Post-Treatment | 14.8375 [3.152 to 26.523]

4. Secondary Outcome: Albumin Level
Description: Pre and Post levels.
Time Frame: 6 months
Population: Only 2 subjects completed the study. Further analysis was not done because power was not met.
Measure: Mean (Full Range); unit: g/dL
Arm/Group | Treatment Group (One Arm Only Study)
Number analyzed (Participants) | 2
g/dL
  Average Pre-Treatment | 3.9 [3.9 to 3.9]
  Average Post-Treatment | 4.05 [3.8 to 4.3]

5. Secondary Outcome: ESA (Erythorpoietic Stimulating Agent) Dose Requirement
Description: Comparison of the average ESA dose used in the 3 month before and the last 3 months of the study.
Time Frame: 6 months
Population: Data for this outcome measure was not collected.
Arm/Group | Treatment Group (One Arm Only Study)
Number analyzed (Participants) | 0
Value | 0

6. Secondary Outcome: Hemoglobin Level
Description: Pre and Post Levels
Time Frame: 6 months
Population: Only 2 subjects completed the study. Further analysis was not done because power was not met.
Measure: Mean (Full Range); unit: g/dL
Arm/Group | Treatment Group (One Arm Only Study)
Number analyzed (Participants) | 2
g/dL
  Average Pre-Treatment | 11.6 [10.9 to 12.3]
  Average Post-Treatment | 10.15 [9.3 to 11]

7. Secondary Outcome: Rate of Cardiovascular Events
Description: Comparison of the average major cardiovascular events (myocardial infarction and/or stroke) in the 3 month before and the last 3 months of the study.
Time Frame: 6 months
Population: Data for this outcome measure was not collected from the medical record due to early termination of the study.
Arm/Group | Treatment Group (One Arm Only Study)
Number analyzed (Participants) | 0
Value | 0

8. Secondary Outcome: Hemodialysis Access Stenosis/Thrombosis
Description: Comparison of the average hemodialysis access stenosis/thrombosis requiring intervention in the 3 month before and the last 3 months of the study.
Time Frame: 6 months
Population: Data for this outcome measure was not collected from the medical record due to early termination of the study.
Arm/Group | Treatment Group (One Arm Only Study)
Number analyzed (Participants) | 0
Value | 0

9. Secondary Outcome: Number of Completed Subjects With Significant Increase in ALT (Alanine Aminotransferase).
Description: The number of subjects with significant rise in ALT but not to the extent requiring removal from the study (rise to more than 3 times the upper limit of the normal range)
Time Frame: 6 months (checked monthly)
Measure: Number; unit: Participants
Arm/Group | Treatment Group (One Arm Only Study)
Number analyzed (Participants) | 2
Participants | 0

ADVERSE EVENTS:
Time Frame: 6 months (the time between the first and the second scan)
Arm/Group | Treatment Group (One Arm Only Study)
Serious Adverse Events (participants affected / at risk) | 1/22
Other Adverse Events (participants affected / at risk) | 2/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (One Arm Only Study) (N=22)
Atrial Fibrillation (Cardiac disorders) | 1 (1) — One subject with pre-existing atrial fibrillation developed another episode of atrial fibrillation and was taken off the study out of abundance of caution and was reported to IRB.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (One Arm Only Study) (N=22)
Flushing (Skin and subcutaneous tissue disorders) | 2 (2)
GI upset (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes